CLINICAL TRIAL: NCT06928844
Title: Role of Low Dose Injectable Progesterone in Triggering Ovulation: A Randomized Controlled Trial
Brief Title: Role of Low Dose Injectable Progesterone in Triggering Ovulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The General Authority for Teaching Hospitals and Institutes (Network)
Responsible Party: Principal Investigator, Abeer Ali Elshabacy, Assistant Scientific Consultant Obstetrics and Gynecology Benha Teaching Hospital, The General Authority for Teaching Hospitals and Institutes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1017/12/24
Record Dates: First submitted 2025-02-12; First posted 2025-04-15 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Low Dose; Progesterone; Triggering Ovulation
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progesterone group (Experimental): Women will receive low dose progesterone 5 mg intramuscularly as a study group.
  Interventions: Drug: Progesterone
- Control group (Placebo Comparator): Women will receive placebo as a control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — Women will receive low dose progesterone 5 mg intramuscularly as a study group. (Letrozole 2.5 mg/day will be given from cycle day 3 onwards for only 5 days).
  Arms: Progesterone group
Drug: Placebo — Women will receive placebo as a control group. (Placebo 2.5 mg/day will be given from cycle day 3 onwards for only 5 days).
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the role of low dose injectable progesterone in triggering ovulation.

DETAILED DESCRIPTION:
Infertility affects approximately 10-15% of couples attempting pregnancy, with no readily identifiable cause found in 15-30% of these patients, resulting in a diagnosis of unexplained infertility.

Kol and Itskovitz-Eldor stated that when using GnRH agonist to trigger ovulation in IVF cycles, the LH surge is associated with a rapid rise of progesterone and the attainment of peak E2 levels through the first 12 h after GnRH agonist administration which is followed by a temporary suppression of progesterone biosynthesis and a gradual drop in E2 levels during the 24 h before follicle aspiration. After oocyte retrieval, a second rise in progesterone and continuous fall in E2 are noted, reflecting transitions from follicular to luteal phase in ovarian steroidogenesis.

Letrozole (LE) is a nonsteroidal, highly selective oral aromatase inhibitor (AI) that inhibits the synthesis of oestrogen and increases the secretion of endogenous gonadotropin by diminishing negative feedback to stimulate ovulation. Currently, letrozole is widely used as an adjunct for IVF cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 35 years.
* Infertile women.
* Basal follicle-stimulating hormone (FSH) level <10 mIU/ml.

Exclusion Criteria:

* Poor ovarian reserve.
* Immunological disease.
* Endometriosis.
* Uterine abnormality.
* Body mass index (BMI) >30 kg/m2.
* Endometrial thickness <8 or >12 mm on the day of triggering.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile women
Enrollment: 120 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of ovulation rates | 10-12 days of the menstrual cycle
  Incidence of ovulation rates will be recorded.

SECONDARY OUTCOMES:
Follicle stimulating hormone (FSH)levels | 10-12 days of the menstrual cycle
  Follicle stimulating hormone (FSH) will be measured on day 3, day 8-10 and day 10-12 of the menstrual cycle, as well as the day of trigger and oocyte retrieval.
Luteinizing hormone (LH)levels | 10-12 days of the menstrual cycle
  Luteinizing hormone (LH) will be measured on day 3, day 8-10 and day 10-12 of the menstrual cycle, as well as the day of trigger and oocyte retrieval).
Estradiol (E2) levels | 10-12 days of the menstrual cycle
  Estradiol (E2) will be measured on day 3, day 8-10 and day 10-12 of the menstrual cycle, as well as the day of trigger and oocyte retrieval.
Progesterone levels | 10-12 days of the menstrual cycle
  Progesterone levels will be measured on day 3, day 8-10 and day 10-12 of the menstrual cycle, as well as the day of trigger and oocyte retrieval.
Number of oocytes | 8 days of the menstrual cycle
  Number of oocytes will be recorded. Ovulation monitoring will be done from the last day of the cycle until ovulation occurs approximately in the middle of the cycle.
Mature oocytes | 16 days of the menstrual cycle
  Mature oocytes will be recorded.
Clinical pregnancy rate. | One week late from the previous menstrual cycle
  Clinical pregnancy rate will be recorded.
Biochemical pregnancy | 16 days of the menstrual cycle
  Biochemical pregnancy will be recorded through a blood pregnancy test on the date of the next menstrual period
Early miscarriage rate | 16 days of the menstrual cycle
  Early miscarriage rate will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Teaching Hospitals and Institutes, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.